CLINICAL TRIAL: NCT01003483
Title: Orlistat Administration Facilitates the Obesity Treatment Among Obese PCOS Women
Brief Title: Metformin Versus Orlistat in Obese Polycystic Ovary Syndrome (PCOS) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yazd Research & Clinical Center for Infertility (Other)
Collaborators: Yazd Medical University (Other)
Responsible Party: Principal Investigator, Nasim Tabibnejad, Dr., Yazd Research & Clinical Center for Infertility
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 616
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Obesity
Keywords: metformin; orlistat; pcos; obese
MeSH Terms: conditions — Obesity; Polycystic Ovary Syndrome | interventions — Orlistat

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orlistat (Experimental): The dose of 120 mg orlistat was taken three times daily and the dose remained constant throughout the study period.
  Interventions: Drug: orlistat
- Metformin (Experimental): The dose of metformin was increased step - wise, from 500 mg once daily for the first week to 500 mg twice daily for the next week, and to 500 mg three times daily for the remaining study period .
  Interventions: Drug: orlistat

INTERVENTIONS:
Drug: orlistat — Tablet,120mg,three times a day,three months
  Other Names: Xenical

SUMMARY:
The purpose of this study is to compare the influence of Orlistat and Metformin on obesity treatment in obese PCOS women.

DETAILED DESCRIPTION:
In a randomized clinical trial study, 80 obese women with BMI≥30, oligomenorrhae, hirsutism and presence of > 12 ovarian follicles (2-10mm diameter), were evaluated. In metformin group , metformin was administered for patients 1500 mg daily for three months. In orlistate group, patients used orlistat tablets (120 mg, 3 times a day) for three months. BMI, serum LH and FSH levels, serum triglyceride and cholesterol levels and also patients' ovulation was compared before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* BMI>= 30
* PCOS

Exclusion Criteria:

* Drug use during last three months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2008-12-01 (Actual); Primary Completion 2009-08 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 3 months

SECONDARY OUTCOMES:
Ovulatory | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Abbas Aflatoonian, Professor, Principal Investigator — Research and Clinical center for Infertility
Locations (1):
- Research and Clinical Center for Infertility, Yazd, Iran